CLINICAL TRIAL: NCT02509702
Title: Text Messages to Increase Attendance to Follow-up Cervical Cancer Screening Appointments Among HPV Positive Tanzanian Women (Connected2Care)
Brief Title: Use of SMSs to Improve Attendance to Cervical Cancer Follow-up Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marianne Andersen (Other)
Responsible Party: Sponsor-Investigator, Marianne Andersen, Clinical professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Connected2Care
Record Dates: First submitted 2015-06-15; First posted 2015-07-28 (Estimated); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Cervical Cancer
Keywords: Mobile health; Screening; Early detection of cancer; HPV; SMS intervention; RCT; Tanzania
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connected to Care (Experimental): The SMS intervention will consist of 15 text messages that will be sent to the intervention group over a period of 10 months. There will be two types of text messages: (1) educational text messages; and (2) SMS reminders for the follow-up appointment.
  Interventions: Behavioral: Connected to Care
- Control (No Intervention): The control group will receive standard care, which is a follow-up appointment at 14 months written on an appointment card.

INTERVENTIONS:
Behavioral: Connected to Care — 10 health educative SMSs' sent once a month 5 SMS-reminders for follow-up appointment sent on days -14, -7, -1 pre- follow-up appointment, and +1, +7 post follow-up appointment
  Arms: Connected to Care

SUMMARY:
This study evaluates the effect of the SMS intervention 'Connected2Care' on the attendance rate to cervical cancer screening follow-up appointments.

DETAILED DESCRIPTION:
Connected2Care is a non-blinded, multicentre, parallel-group, randomised controlled trial. Tanzanian Women testing positive to HR HPV at inclusion are randomly assigned in an allocation ratio of 1:1 to the SMS intervention or the control group (standard care). In a period of 10 months, the intervention group will receive 15 one-directional health educative text messages and SMS-reminders for their appointment. The total sample size will be 700 with 350 women in each study arm. Primary outcome is attendance rate for follow-up. Secondary objectives are cost-effectiveness measured through incremental ratios and knowledge of cervical cancer by a 16-item true/false scale questionnaire at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* HPV positive
* Age 25 - 60 years
* Private mobile phone

Exclusion Criteria:

* Pregnant on day of enrolment
* Menstruating on day of enrolment
* Hysterectomy
* Diagnosed with cervical pre-cancer within past 12 months
* Diagnosed with cervical cancer
* Invalid mobile phone number
* Unreachable when trying to convey HPV positive result

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 705 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Effect of SMS intervention on attendance rate to follow-up screening appointment | up to 14 months
  The effect measure of the intervention is the 14-month follow-up attendance rate for HPV positive women. The number of women in the intervention group that attend follow-up screening will be compared to the the number of women that attend follow-up screening in the control group.

SECONDARY OUTCOMES:
Acceptability of text message intervention | Baseline + 2 years Follow-up (likert scale)
  6-point Likert scale (1: I do not like it at all - 6: I like it very much)
Acceptability of text message intervention | 2 years
  Qualitative interviews. Open-ended

OTHER OUTCOMES:
Cost-effectiveness of intervention | Baseline + 14 months
  Incremental cost-effectiveness ratio
Knowledge of cervical cancer and screening | Baselie + 14 months
  16 item true-false questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Rasch, MD, Study Chair — University of Southern Denmark; Julius Mwaiselage, MD, Study Chair — Ocean Road Cancer Institute
Locations (3):
- Tanzania (3):
  - Mawenzi Regional Referral Hospital, Moshi, Kilimanjaro
  - Ocean Road Cancer Institute (ORCI), Dar es Salaam
  - Kilimanjaro Christian Medical Centre (KCMC), Moshi

REFERENCES:
- [Background] Linde DS, Andersen MS, Mwaiselage JD, Manongi R, Kjaer SK, Rasch V. Text messages to increase attendance to follow-up cervical cancer screening appointments among HPV-positive Tanzanian women (Connected2Care): study protocol for a randomised controlled trial. Trials. 2017 Nov 21;18(1):555. doi: 10.1186/s13063-017-2215-x. PMID 29162148
- [Derived] Lokke KF, Rasch V, Mwaiselage J, Gammeltoft T, Linde DS. Acceptability of text messages and knowledge change for cervical cancer screening: a Tanzanian mixed methods study. BMJ Open. 2022 Sep 19;12(9):e058450. doi: 10.1136/bmjopen-2021-058450. PMID 36123109
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Linde DS, Andersen MS, Mwaiselage J, Manongi R, Kjaer SK, Rasch V. Effectiveness of One-Way Text Messaging on Attendance to Follow-Up Cervical Cancer Screening Among Human Papillomavirus-Positive Tanzanian Women (Connected2Care): Parallel-Group Randomized Controlled Trial. J Med Internet Res. 2020 Apr 2;22(4):e15863. doi: 10.2196/15863. PMID 32238335
- [Derived] Linde DS, Rasch V, Mwaiselage JD, Gammeltoft TM. Competing needs: a qualitative study of cervical cancer screening attendance among HPV-positive women in Tanzania. BMJ Open. 2019 Feb 27;9(2):e024011. doi: 10.1136/bmjopen-2018-024011. PMID 30819704